CLINICAL TRIAL: NCT05275608
Title: Effects of Very Low Calorie Ketogenic Diet on Microbiota, Adipose Tissue and Immunitary Regulation: Pilot Study on Patients with Metabolic Syndrome
Brief Title: Effects of VLCKD in Metabolic Syndrome
Acronym: KETO-MI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero Universitaria Maggiore della Carita (Other)
Collaborators: Laboratoire THERASCIENCE (Unknown)
Responsible Party: Principal Investigator, Flavia Prodam, Associated Prof. in Clinical Nutrition and MD, Azienda Ospedaliero Universitaria Maggiore della Carita
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CE 296/21
Record Dates: First submitted 2022-02-21; First posted 2022-03-11 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Diabetes Mellitus, Type 2; Non-alcoholic Fatty Liver Disease; Obesity; Metabolic Syndrome
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Non-alcoholic Fatty Liver Disease; Obesity; Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- VLCKD (Experimental): 20 Patients recruited from our endocrinology department that will keep the same medical visits frequency and drugs and accept to be randomized to one of the two groups.
  Inclusion criteria:
  * Age 25-65
  * BMI 30-40 mg/m2
  * NAFLD
  * DM2 drug-treated (metformin, SGLT2 inhibitors, GLP-1 analogues, DPPIV inhibitors, insulin) and HbA1c > 7 and < 10 %.
  Interventions: Dietary Supplement: VLCKD diet with replacing meals
- Hypocaloric Mediterranean Diet (Active Comparator): 20 Patients recruited from our endocrinology department that will keep the same medical visits frequency and drugs and accept to be randomized to one of the two groups.
  Inclusion criteria:
  * Age 25-65
  * BMI 30-40 mg/m2
  * NAFLD
  * DM2 drug-treated (metformin, SGLT2 inhibitors, GLP-1 analogues, DPPIV inhibitors, insulin) and HbA1c > 7 and < 10 %.
  Interventions: Behavioral: Hypocaloric mediterranean Diet

INTERVENTIONS:
Dietary Supplement: VLCKD diet with replacing meals — Patients will receive an accurate teaching + brochure on VLCKD diet from an expert dietician and freely receive the correct amount of supplements provided from Labotaoire Therascience (4 or 5 meals). The supplements contain (in total) between 600 and 800 kcal, mainly fats, 1,2/1,5 g/body weight of proteins, very low amount of charbohydrates (<30/40g/die), 10-20g fibers, + minerals and vitamins covering the needings of patients. After 6-8 weeks, 1 meal will be replaced with a natural dish rich in proteins.
  Arms: VLCKD
Behavioral: Hypocaloric mediterranean Diet — Patients will receive an accurate teaching + brochure on an hypocaloric Mediterranean style diet (LARN 2014) from an expert dietician. Patients will follow the istructions on grams and foods to eat. The calories will be around minus 400-500 kcal from energy requirement (measured by indirect calorimetry * physical activity score).
  Arms: Hypocaloric Mediterranean Diet

SUMMARY:
VLCKD has showed to be an impactful diet on several metabolism aspects and has proven to be useful for preventing and treating diabetes mellitus type 2, overweight, chronic inflammation and fatty liver.

For this reason, the aim of this pilot study is to examinate the potential effect of a VLCKD on a group of patients that contemporarily have DM2, obesity and Non alcholic fatty liver disease (NAFLD), comparing the results with an ipocaloric diet based on Mediterranean Principles and Italian LARN (SINU 2014).

This study will consider several interrelated outcomes such as anthropometric data, hematochemical and hormonal parameters, questionnaires, stool microbiota and omics, blood microvescicles, urine tests, instrumental tests (DXA, BIVA, ecographies), biopses and functional tests.

40 subjects will be evaluated and divided in two groups of 20 (VLCKD) and 20 (MedDiet).

ELIGIBILITY:
Inclusion Criteria:

* Age 25-65
* BMI 30-40 mg/m2
* NAFLD
* DM2 drug-treated (metformin, SGLT2 inhibitors, GLP-1 analogues, DPPIV inhibitors, basal insulin) and HbA1c > 7 and < 10 %.

Exclusion Criteria:

* Secondary obesity due to genetic or endocrinologic causes.
* renal disease with eGFR < 45 mL/min/1.73m2 or macroalbuminuria or calculosis
* insulin basal + bolus or HbA1c% >10.0%
* Other types of DM
* ipopituitarism or adrenal insufficiency
* antibiotics use less than 3 months before the first visit

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-11-07 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in weight | Change from Baseline BMI at 15 days, 30 days, 60 days, 90 days
  Variation of body weight assessed through body mass index change (BMI)(kg/m2)
Change in body circumferences | Change from Baseline circumferences at 15 days, 30 days, 60 days, 90 days
  Variation of body circumferences (waist, hips)
Change in metabolic control | Change from Baseline blood glucose at 15 days, 30 days, 60 days, 90 days
  Variation of blood glucose
Change in metabolic control | Change from Baseline lipid profile at 15 days, 30 days, 60 days, 90 days
  Change of cardio-metabolic risk factors: lipid profile

SECONDARY OUTCOMES:
Change in Metabolic control | Change from Baseline HOMA-IR at 15 days, 30 days, 60 days, 90 days
  Change of cardio-metabolic risk factors: insulin resistance (HOMA-IR)
Change in kidney profile | Change from Baseline Serum Creatinin at 15 days, 30 days, 60 days, 90 days
  Variation of serum creatinin
Change in liver profile | Change from Baseline liver profile at 15 days, 30 days, 60 days, 90 days
  Variation of liver profile (AST, ALT, GGT, bilirubin)
Change in uric acid | Change from Baseline uric acid at 15 days, 30 days, 60 days, 90 days
  Variation of uric acid in blood
Change in blood pressure | Change from Baseline blood pressure at 15 days, 30 days, 60 days, 90 days
  Variation of blood pressure (diastolic and sistolic)
Change in body composition | Change from Baseline fat mass% at 15 days, 30 days, 60 days, 90 days
  Change of body composition (fat mass %) (BIVA)
Change in body composition | Change from Baseline fat mass% at 90 days
  Change of body composition (fat mass %) (DXA)
Change in muscolar functionality | Change from Baseline scores at 30, 90 days
  Changes observed from functional tests (handgrip strenght)
Change in muscolar functionality | Change from Baseline scores at 30, 90 days
  Changes observed from functional tests (short physical portable battery score)
Change in muscolar functionality | Change from Baseline scores at 30, 90 days
  Changes observed from functional tests (time up and go test)
Change in hormones | Change from Baseline blood hormones at 15, 30 days, 60 days, 90 days
  Variation of hormones in blood (ghrelin, leptin, adiponectin)
Change in hormones | Change from Baseline blood hormones at 15, 30 days, 60 days, 90 days
  Variation of hormones in blood (irisin)
Change in hormones | Change from Baseline blood hormones at 15, 30 days, 60 days, 90 days
  Variation of hormones in blood (zonulin)
Change in hormones | Change from Baseline blood hormones at 15, 30 days, 60 days, 90 days
  Variation of hormones in blood (asprosin)
Change in hormones | Change from Baseline blood hormones at 15, 30 days, 60 days, 90 days
  Variation of hormones in blood (TSH)
Change in hormones | Change from Baseline blood hormones at 15, 30 days, 60 days, 90 days
  Variation of hormones in blood (FT4)
Change in hormones | Change from Baseline blood hormones at 15, 30 days, 60 days, 90 days
  Variation of hormones in blood (PTH)
Change in hormones | Change from Baseline blood hormones at 15, 30 days, 60 days, 90 days
  Variation of hormones in blood (25OH vitamin D)
Change in hormones | Change from Baseline blood hormones at 15, 30 days, 60 days, 90 days
  Variation of hormones in blood (PYY)
Change in hormones | Change from Baseline blood hormones at 15, 30 days, 60 days, 90 days
  Variation of hormones in blood (IGF-1)
Change in blood ketones | Change from Baseline blood ketones at 15, 30 days, 60 days, 90 days
  Variation of ketones in blood
Change in basal metabolic rate | Change from Baseline basal metabolic rate at 90 days
  Variation of basal metabolic rate through indirect calorimetry
Change in urine ketones | Change from Baseline urine ketones at 15, 30 days, 60 days, 90 days
  Variation of urine excretion in terms of ketones
Change in urine nitrogen excretion | Change from Baseline urine nitrogen at 15, 30 days, 60 days, 90 days
  Variation of urine excretion in terms of nitrogen
Change in omics profile | Change from Baseline omic profile of stools at 15, 30 days, 60 days, 90 days
  Variation of metabolomic profile of stools through liquid and gas chromatography
Change in omics profile | Change from Baseline omic profile of stools at 15, 30 days, 60 days, 90 days
  Variation of lipidomic profile of stools through liquid and gas chromatography
Change in omics profile | Change from Baseline omic profile of stools at 15, 30 days, 60 days, 90 days
  Variation of proteomic profile of stools through liquid and gas chromatography
Change in microbiota | Change from Baseline of prevalence of microbiota phyla at 15, 30 days, 60 days, 90 days
  Variation of prevalence of microbiota phyla through DNA sequencing of stools
Change in inflammatory status | Change from Baseline CRP and cytokines at 15, 30 days, 60 days, 90 days
  Variation of inflammatory status in blood (C-reactive protein CRP)
Change in inflammatory status | Change from Baseline cytokines at 15, 30 days, 60 days, 90 days
  Variation of inflammatory status in blood (cytokines count)

CONTACTS AND LOCATIONS:
Locations (1):
- : Italy Pediatric Endocrine Service of AOU Maggiore della Carità of Novara; SCDU of Pediatrics, Department of Health Sciences, University of Eastern Piedmont, Novara, Italy, Italy

REFERENCES:
- [Background] Abbasi J. Interest in the Ketogenic Diet Grows for Weight Loss and Type 2 Diabetes. JAMA. 2018 Jan 16;319(3):215-217. doi: 10.1001/jama.2017.20639. No abstract available. PMID 29340675
- [Background] American Diabetes Association. 5. Lifestyle Management: Standards of Medical Care in Diabetes-2019. Diabetes Care. 2019 Jan;42(Suppl 1):S46-S60. doi: 10.2337/dc19-S005. PMID 30559231
- [Background] American Diabetes Association. 8. Obesity Management for the Treatment of Type 2 Diabetes: Standards of Medical Care in Diabetes-2019. Diabetes Care. 2019 Jan;42(Suppl 1):S81-S89. doi: 10.2337/dc19-S008. PMID 30559234
- [Background] Ang QY, Alexander M, Newman JC, Tian Y, Cai J, Upadhyay V, Turnbaugh JA, Verdin E, Hall KD, Leibel RL, Ravussin E, Rosenbaum M, Patterson AD, Turnbaugh PJ. Ketogenic Diets Alter the Gut Microbiome Resulting in Decreased Intestinal Th17 Cells. Cell. 2020 Jun 11;181(6):1263-1275.e16. doi: 10.1016/j.cell.2020.04.027. Epub 2020 May 20. PMID 32437658
- [Background] Very low-calorie diets. National Task Force on the Prevention and Treatment of Obesity, National Institutes of Health. JAMA. 1993 Aug 25;270(8):967-74. PMID 8345648
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Background] Baker ST, Jerums G, Prendergast LA, Panagiotopoulos S, Strauss BJ, Proietto J. Less fat reduction per unit weight loss in type 2 diabetic compared with nondiabetic obese individuals completing a very-low-calorie diet program. Metabolism. 2012 Jun;61(6):873-82. doi: 10.1016/j.metabol.2011.10.017. Epub 2011 Dec 5. PMID 22146094
- [Background] Barengolts E. GUT MICROBIOTA, PREBIOTICS, PROBIOTICS, AND SYNBIOTICS IN MANAGEMENT OF OBESITY AND PREDIABETES: REVIEW OF RANDOMIZED CONTROLLED TRIALS. Endocr Pract. 2016 Oct;22(10):1224-1234. doi: 10.4158/EP151157.RA. Epub 2016 Jul 13. PMID 27409822
- [Background] Depommier C, Everard A, Druart C, Plovier H, Van Hul M, Vieira-Silva S, Falony G, Raes J, Maiter D, Delzenne NM, de Barsy M, Loumaye A, Hermans MP, Thissen JP, de Vos WM, Cani PD. Supplementation with Akkermansia muciniphila in overweight and obese human volunteers: a proof-of-concept exploratory study. Nat Med. 2019 Jul;25(7):1096-1103. doi: 10.1038/s41591-019-0495-2. Epub 2019 Jul 1. PMID 31263284
- [Background] Cabrera-Mulero A, Tinahones A, Bandera B, Moreno-Indias I, Macias-Gonzalez M, Tinahones FJ. Keto microbiota: A powerful contributor to host disease recovery. Rev Endocr Metab Disord. 2019 Dec;20(4):415-425. doi: 10.1007/s11154-019-09518-8. PMID 31720986
- [Background] Cappellano G, Morandi EM, Rainer J, Grubwieser P, Heinz K, Wolfram D, Bernhard D, Lobenwein S, Pierer G, Ploner C. Human Macrophages Preferentially Infiltrate the Superficial Adipose Tissue. Int J Mol Sci. 2018 May 8;19(5):1404. doi: 10.3390/ijms19051404. PMID 29738484
- [Background] Caprio M, Infante M, Moriconi E, Armani A, Fabbri A, Mantovani G, Mariani S, Lubrano C, Poggiogalle E, Migliaccio S, Donini LM, Basciani S, Cignarelli A, Conte E, Ceccarini G, Bogazzi F, Cimino L, Condorelli RA, La Vignera S, Calogero AE, Gambineri A, Vignozzi L, Prodam F, Aimaretti G, Linsalata G, Buralli S, Monzani F, Aversa A, Vettor R, Santini F, Vitti P, Gnessi L, Pagotto U, Giorgino F, Colao A, Lenzi A; Cardiovascular Endocrinology Club of the Italian Society of Endocrinology. Very-low-calorie ketogenic diet (VLCKD) in the management of metabolic diseases: systematic review and consensus statement from the Italian Society of Endocrinology (SIE). J Endocrinol Invest. 2019 Nov;42(11):1365-1386. doi: 10.1007/s40618-019-01061-2. Epub 2019 May 20. PMID 31111407
- [Background] Capstick F, Brooks BA, Burns CM, Zilkens RR, Steinbeck KS, Yue DK. Very low calorie diet (VLCD): a useful alternative in the treatment of the obese NIDDM patient. Diabetes Res Clin Pract. 1997 May;36(2):105-11. doi: 10.1016/s0168-8227(97)00038-7. PMID 9229194
- [Background] Caresio C, Salvi M, Molinari F, Meiburger KM, Minetto MA. Fully Automated Muscle Ultrasound Analysis (MUSA): Robust and Accurate Muscle Thickness Measurement. Ultrasound Med Biol. 2017 Jan;43(1):195-205. doi: 10.1016/j.ultrasmedbio.2016.08.032. Epub 2016 Oct 6. PMID 27720522
- [Background] Cicero AF, Benelli M, Brancaleoni M, Dainelli G, Merlini D, Negri R. Middle and Long-Term Impact of a Very Low-Carbohydrate Ketogenic Diet on Cardiometabolic Factors: A Multi-Center, Cross-Sectional, Clinical Study. High Blood Press Cardiovasc Prev. 2015 Dec;22(4):389-94. doi: 10.1007/s40292-015-0096-1. Epub 2015 May 19. PMID 25986079
- [Background] Cunha GM, Guzman G, Correa De Mello LL, Trein B, Spina L, Bussade I, Marques Prata J, Sajoux I, Countinho W. Efficacy of a 2-Month Very Low-Calorie Ketogenic Diet (VLCKD) Compared to a Standard Low-Calorie Diet in Reducing Visceral and Liver Fat Accumulation in Patients With Obesity. Front Endocrinol (Lausanne). 2020 Sep 14;11:607. doi: 10.3389/fendo.2020.00607. eCollection 2020. PMID 33042004
- [Background] David LA, Maurice CF, Carmody RN, Gootenberg DB, Button JE, Wolfe BE, Ling AV, Devlin AS, Varma Y, Fischbach MA, Biddinger SB, Dutton RJ, Turnbaugh PJ. Diet rapidly and reproducibly alters the human gut microbiome. Nature. 2014 Jan 23;505(7484):559-63. doi: 10.1038/nature12820. Epub 2013 Dec 11. PMID 24336217
- [Background] Daien CI, Pinget GV, Tan JK, Macia L. Detrimental Impact of Microbiota-Accessible Carbohydrate-Deprived Diet on Gut and Immune Homeostasis: An Overview. Front Immunol. 2017 May 12;8:548. doi: 10.3389/fimmu.2017.00548. eCollection 2017. PMID 28553291
- [Background] Dehghan M, Mente A, Zhang X, Swaminathan S, Li W, Mohan V, Iqbal R, Kumar R, Wentzel-Viljoen E, Rosengren A, Amma LI, Avezum A, Chifamba J, Diaz R, Khatib R, Lear S, Lopez-Jaramillo P, Liu X, Gupta R, Mohammadifard N, Gao N, Oguz A, Ramli AS, Seron P, Sun Y, Szuba A, Tsolekile L, Wielgosz A, Yusuf R, Hussein Yusufali A, Teo KK, Rangarajan S, Dagenais G, Bangdiwala SI, Islam S, Anand SS, Yusuf S; Prospective Urban Rural Epidemiology (PURE) study investigators. Associations of fats and carbohydrate intake with cardiovascular disease and mortality in 18 countries from five continents (PURE): a prospective cohort study. Lancet. 2017 Nov 4;390(10107):2050-2062. doi: 10.1016/S0140-6736(17)32252-3. Epub 2017 Aug 29. PMID 28864332
- [Background] Di Rosa C, Lattanzi G, Taylor SF, Manfrini S, Khazrai YM. Very low calorie ketogenic diets in overweight and obesity treatment: Effects on anthropometric parameters, body composition, satiety, lipid profile and microbiota. Obes Res Clin Pract. 2020 Nov-Dec;14(6):491-503. doi: 10.1016/j.orcp.2020.08.009. Epub 2020 Sep 9. PMID 32919928
- [Background] Estruch R, Martinez-Gonzalez MA, Corella D, Salas-Salvado J, Ruiz-Gutierrez V, Covas MI, Fiol M, Gomez-Gracia E, Lopez-Sabater MC, Vinyoles E, Aros F, Conde M, Lahoz C, Lapetra J, Saez G, Ros E; PREDIMED Study Investigators. Effects of a Mediterranean-style diet on cardiovascular risk factors: a randomized trial. Ann Intern Med. 2006 Jul 4;145(1):1-11. doi: 10.7326/0003-4819-145-1-200607040-00004. PMID 16818923
- [Background] Gregg EW, Shaw JE. Global Health Effects of Overweight and Obesity. N Engl J Med. 2017 Jul 6;377(1):80-81. doi: 10.1056/NEJMe1706095. Epub 2017 Jun 12. No abstract available. PMID 28604226
- [Background] Goday A, Bellido D, Sajoux I, Crujeiras AB, Burguera B, Garcia-Luna PP, Oleaga A, Moreno B, Casanueva FF. Short-term safety, tolerability and efficacy of a very low-calorie-ketogenic diet interventional weight loss program versus hypocaloric diet in patients with type 2 diabetes mellitus. Nutr Diabetes. 2016 Sep 19;6(9):e230. doi: 10.1038/nutd.2016.36. PMID 27643725
- [Background] Gu Y, Yu H, Li Y, Ma X, Lu J, Yu W, Xiao Y, Bao Y, Jia W. Beneficial effects of an 8-week, very low carbohydrate diet intervention on obese subjects. Evid Based Complement Alternat Med. 2013;2013:760804. doi: 10.1155/2013/760804. Epub 2013 Mar 14. PMID 23573151
- [Background] Guralnik JM, Ferrucci L, Simonsick EM, Salive ME, Wallace RB. Lower-extremity function in persons over the age of 70 years as a predictor of subsequent disability. N Engl J Med. 1995 Mar 2;332(9):556-61. doi: 10.1056/NEJM199503023320902. PMID 7838189
- [Background] Heinsen FA, Fangmann D, Muller N, Schulte DM, Ruhlemann MC, Turk K, Settgast U, Lieb W, Baines JF, Schreiber S, Franke A, Laudes M. Beneficial Effects of a Dietary Weight Loss Intervention on Human Gut Microbiome Diversity and Metabolism Are Not Sustained during Weight Maintenance. Obes Facts. 2016;9(6):379-391. doi: 10.1159/000449506. Epub 2016 Nov 30. PMID 27898428
- [Background] Invernizzi M, Rizzi M, Carda S, Cisari C, Molinari C, Reno F. Mini invasive skeletal muscle biopsy technique with a tri-axial end cut needle. Eur Rev Med Pharmacol Sci. 2015 Jul;19(13):2446-51. PMID 26214781
- [Background] Jensen MD, Ryan DH, Apovian CM, Ard JD, Comuzzie AG, Donato KA, Hu FB, Hubbard VS, Jakicic JM, Kushner RF, Loria CM, Millen BE, Nonas CA, Pi-Sunyer FX, Stevens J, Stevens VJ, Wadden TA, Wolfe BM, Yanovski SZ; American College of Cardiology/American Heart Association Task Force on Practice Guidelines; Obesity Society. 2013 AHA/ACC/TOS guideline for the management of overweight and obesity in adults: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines and The Obesity Society. J Am Coll Cardiol. 2014 Jul 1;63(25 Pt B):2985-3023. doi: 10.1016/j.jacc.2013.11.004. Epub 2013 Nov 12. No abstract available. PMID 24239920
- [Background] Kipnis V, Midthune D, Freedman L, Bingham S, Day NE, Riboli E, Ferrari P, Carroll RJ. Bias in dietary-report instruments and its implications for nutritional epidemiology. Public Health Nutr. 2002 Dec;5(6A):915-23. doi: 10.1079/PHN2002383. PMID 12633516
- [Background] Laurans L, Venteclef N, Haddad Y, Chajadine M, Alzaid F, Metghalchi S, Sovran B, Denis RGP, Dairou J, Cardellini M, Moreno-Navarrete JM, Straub M, Jegou S, McQuitty C, Viel T, Esposito B, Tavitian B, Callebert J, Luquet SH, Federici M, Fernandez-Real JM, Burcelin R, Launay JM, Tedgui A, Mallat Z, Sokol H, Taleb S. Genetic deficiency of indoleamine 2,3-dioxygenase promotes gut microbiota-mediated metabolic health. Nat Med. 2018 Aug;24(8):1113-1120. doi: 10.1038/s41591-018-0060-4. Epub 2018 Jun 25. PMID 29942089
- [Background] Lee MJ, Pickering RT, Puri V. Prolonged efficiency of siRNA-mediated gene silencing in primary cultures of human preadipocytes and adipocytes. Obesity (Silver Spring). 2014 Apr;22(4):1064-9. doi: 10.1002/oby.20641. Epub 2013 Dec 5. PMID 24307633
- [Background] Li Y, Luo W, Deng Z, Lei G. Diet-Intestinal Microbiota Axis in Osteoarthritis: A Possible Role. Mediators Inflamm. 2016;2016:3495173. doi: 10.1155/2016/3495173. Epub 2016 Aug 17. PMID 27610004
- [Background] Lim EL, Hollingsworth KG, Aribisala BS, Chen MJ, Mathers JC, Taylor R. Reversal of type 2 diabetes: normalisation of beta cell function in association with decreased pancreas and liver triacylglycerol. Diabetologia. 2011 Oct;54(10):2506-14. doi: 10.1007/s00125-011-2204-7. Epub 2011 Jun 9. PMID 21656330
- [Background] Malandrucco I, Pasqualetti P, Giordani I, Manfellotto D, De Marco F, Alegiani F, Sidoti AM, Picconi F, Di Flaviani A, Frajese G, Bonadonna RC, Frontoni S. Very-low-calorie diet: a quick therapeutic tool to improve beta cell function in morbidly obese patients with type 2 diabetes. Am J Clin Nutr. 2012 Mar;95(3):609-13. doi: 10.3945/ajcn.111.023697. Epub 2012 Feb 8. PMID 22318758
- [Background] Manfredi M, Conte E, Barberis E, Buzzi A, Robotti E, Caneparo V, Cecconi D, Brandi J, Vanni E, Finocchiaro M, Astegiano M, Gariglio M, Marengo E, De Andrea M. Integrated serum proteins and fatty acids analysis for putative biomarker discovery in inflammatory bowel disease. J Proteomics. 2019 Mar 20;195:138-149. doi: 10.1016/j.jprot.2018.10.017. Epub 2018 Nov 2. PMID 30391485
- [Background] McAllan L, Skuse P, Cotter PD, O'Connor P, Cryan JF, Ross RP, Fitzgerald G, Roche HM, Nilaweera KN. Protein quality and the protein to carbohydrate ratio within a high fat diet influences energy balance and the gut microbiota in C57BL/6J mice. PLoS One. 2014 Feb 10;9(2):e88904. doi: 10.1371/journal.pone.0088904. eCollection 2014. PMID 24520424
- [Background] Meidenbauer JJ, Mukherjee P, Seyfried TN. The glucose ketone index calculator: a simple tool to monitor therapeutic efficacy for metabolic management of brain cancer. Nutr Metab (Lond). 2015 Mar 11;12:12. doi: 10.1186/s12986-015-0009-2. eCollection 2015. PMID 25798181
- [Background] Meijer K, de Vries M, Al-Lahham S, Bruinenberg M, Weening D, Dijkstra M, Kloosterhuis N, van der Leij RJ, van der Want H, Kroesen BJ, Vonk R, Rezaee F. Human primary adipocytes exhibit immune cell function: adipocytes prime inflammation independent of macrophages. PLoS One. 2011 Mar 23;6(3):e17154. doi: 10.1371/journal.pone.0017154. PMID 21448265
- [Background] Monda V, Polito R, Lovino A, Finaldi A, Valenzano A, Nigro E, Corso G, Sessa F, Asmundo A, Nunno ND, Cibelli G, Messina G. Short-Term Physiological Effects of a Very Low-Calorie Ketogenic Diet: Effects on Adiponectin Levels and Inflammatory States. Int J Mol Sci. 2020 May 2;21(9):3228. doi: 10.3390/ijms21093228. PMID 32370212
- [Background] Montesi L, El Ghoch M, Brodosi L, Calugi S, Marchesini G, Dalle Grave R. Long-term weight loss maintenance for obesity: a multidisciplinary approach. Diabetes Metab Syndr Obes. 2016 Feb 26;9:37-46. doi: 10.2147/DMSO.S89836. eCollection 2016. PMID 27013897
- [Background] Moriconi E, Camajani E, Fabbri A, Lenzi A, Caprio M. Very-Low-Calorie Ketogenic Diet as a Safe and Valuable Tool for Long-Term Glycemic Management in Patients with Obesity and Type 2 Diabetes. Nutrients. 2021 Feb 26;13(3):758. doi: 10.3390/nu13030758. PMID 33652834
- [Background] Muscogiuri G, El Ghoch M, Colao A, Hassapidou M, Yumuk V, Busetto L; Obesity Management Task Force (OMTF) of the European Association for the Study of Obesity (EASO). European Guidelines for Obesity Management in Adults with a Very Low-Calorie Ketogenic Diet: A Systematic Review and Meta-Analysis. Obes Facts. 2021;14(2):222-245. doi: 10.1159/000515381. Epub 2021 Apr 21. PMID 33882506
- [Background] Paoli A, Bosco G, Camporesi EM, Mangar D. Ketosis, ketogenic diet and food intake control: a complex relationship. Front Psychol. 2015 Feb 2;6:27. doi: 10.3389/fpsyg.2015.00027. eCollection 2015. PMID 25698989
- [Background] Peisl BYL, Schymanski EL, Wilmes P. Dark matter in host-microbiome metabolomics: Tackling the unknowns-A review. Anal Chim Acta. 2018 Dec 11;1037:13-27. doi: 10.1016/j.aca.2017.12.034. Epub 2017 Dec 30. PMID 30292286
- [Background] Piaggi P, Vinales KL, Basolo A, Santini F, Krakoff J. Energy expenditure in the etiology of human obesity: spendthrift and thrifty metabolic phenotypes and energy-sensing mechanisms. J Endocrinol Invest. 2018 Jan;41(1):83-89. doi: 10.1007/s40618-017-0732-9. Epub 2017 Jul 24. PMID 28741280
- [Background] Podsiadlo D, Richardson S. The timed "Up & Go": a test of basic functional mobility for frail elderly persons. J Am Geriatr Soc. 1991 Feb;39(2):142-8. doi: 10.1111/j.1532-5415.1991.tb01616.x. PMID 1991946
- [Background] Pownall HJ, Bray GA, Wagenknecht LE, Walkup MP, Heshka S, Hubbard VS, Hill J, Kahn SE, Nathan DM, Schwartz AV, Johnson KC; Look AHEAD Research Group. Changes in body composition over 8 years in a randomized trial of a lifestyle intervention: the look AHEAD study. Obesity (Silver Spring). 2015 Mar;23(3):565-72. doi: 10.1002/oby.21005. PMID 25707379
- [Background] Romano L, Marchetti M, Gualtieri P, Di Renzo L, Belcastro M, De Santis GL, Perrone MA, De Lorenzo A. Effects of a Personalized VLCKD on Body Composition and Resting Energy Expenditure in the Reversal of Diabetes to Prevent Complications. Nutrients. 2019 Jul 4;11(7):1526. doi: 10.3390/nu11071526. PMID 31277506
- [Background] Rondanelli M, Gasparri C, Peroni G, Faliva MA, Naso M, Perna S, Bazire P, Sajuox I, Maugeri R, Rigon C. The Potential Roles of Very Low Calorie, Very Low Calorie Ketogenic Diets and Very Low Carbohydrate Diets on the Gut Microbiota Composition. Front Endocrinol (Lausanne). 2021 May 14;12:662591. doi: 10.3389/fendo.2021.662591. eCollection 2021. PMID 34054731
- [Background] Rothberg AE, McEwen LN, Kraftson AT, Fowler CE, Herman WH. Very-low-energy diet for type 2 diabetes: an underutilized therapy? J Diabetes Complications. 2014 Jul-Aug;28(4):506-10. doi: 10.1016/j.jdiacomp.2014.03.014. Epub 2014 Mar 29. PMID 24849710
- [Background] Saslow LR, Daubenmier JJ, Moskowitz JT, Kim S, Murphy EJ, Phinney SD, Ploutz-Snyder R, Goldman V, Cox RM, Mason AE, Moran P, Hecht FM. Twelve-month outcomes of a randomized trial of a moderate-carbohydrate versus very low-carbohydrate diet in overweight adults with type 2 diabetes mellitus or prediabetes. Nutr Diabetes. 2017 Dec 21;7(12):304. doi: 10.1038/s41387-017-0006-9. PMID 29269731
- [Background] Singh RK, Chang HW, Yan D, Lee KM, Ucmak D, Wong K, Abrouk M, Farahnik B, Nakamura M, Zhu TH, Bhutani T, Liao W. Influence of diet on the gut microbiome and implications for human health. J Transl Med. 2017 Apr 8;15(1):73. doi: 10.1186/s12967-017-1175-y. PMID 28388917
- [Background] Steven S, Hollingsworth KG, Al-Mrabeh A, Avery L, Aribisala B, Caslake M, Taylor R. Very Low-Calorie Diet and 6 Months of Weight Stability in Type 2 Diabetes: Pathophysiological Changes in Responders and Nonresponders. Diabetes Care. 2016 May;39(5):808-15. doi: 10.2337/dc15-1942. Epub 2016 Mar 21. PMID 27002059
- [Background] Solito A, Bozzi Cionci N, Calgaro M, Caputo M, Vannini L, Hasballa I, Archero F, Giglione E, Ricotti R, Walker GE, Petri A, Agosti E, Bellomo G, Aimaretti G, Bona G, Bellone S, Amoruso A, Pane M, Di Gioia D, Vitulo N, Prodam F. Supplementation with Bifidobacterium breve BR03 and B632 strains improved insulin sensitivity in children and adolescents with obesity in a cross-over, randomized double-blind placebo-controlled trial. Clin Nutr. 2021 Jul;40(7):4585-4594. doi: 10.1016/j.clnu.2021.06.002. Epub 2021 Jun 11. PMID 34229263
- [Background] Viljanen AP, Lautamaki R, Jarvisalo M, Parkkola R, Huupponen R, Lehtimaki T, Ronnemaa T, Raitakari OT, Iozzo P, Nuutila P. Effects of weight loss on visceral and abdominal subcutaneous adipose tissue blood-flow and insulin-mediated glucose uptake in healthy obese subjects. Ann Med. 2009;41(2):152-60. doi: 10.1080/07853890802446754. PMID 18855190
- [Background] Walker GE, Marzullo P, Prodam F, Bona G, Di Blasio AM. Obesity modifies expression profiles of metabolic markers in superficial and deep subcutaneous abdominal adipose tissue depots. Endocrine. 2014 May;46(1):99-106. doi: 10.1007/s12020-013-0040-x. Epub 2013 Sep 13. PMID 24030694